CLINICAL TRIAL: NCT01759875
Title: Effects of Gastric pH on the Pharmacokinetics of Atazanavir in Healthy Volunteers
Brief Title: Effects of Gastric pH on the Pharmacokinetics of Atazanavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CRS6537
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — Rabeprazole; Betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ritonavir-boosted Atazanavir (Active Comparator)
  Interventions: Drug: Ritonavir-boosted Atazanavir
- Ritonavir-boosted Atazanavir plus Rabeprazole (Experimental)
  Interventions: Drug: Ritonavir-boosted Atazanavir plus Rabeprazole
- Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine HCl (Experimental)
  Interventions: Drug: Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine Hydrochloride

INTERVENTIONS:
Drug: Ritonavir-boosted Atazanavir — Ritonavir (100mg) PO x1 and Atazanavir (300mg) PO x1
  Arms: Ritonavir-boosted Atazanavir
Drug: Ritonavir-boosted Atazanavir plus Rabeprazole — Rabeprazole (20mg) PO twice daily (Days 1-3); Ritonavir (100mg) PO x1 and Atazanavir (300mg) PO x1 (Day 4)
  Arms: Ritonavir-boosted Atazanavir plus Rabeprazole
Drug: Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine Hydrochloride — Rabeprazole (20mg) PO twice daily (Days 1-3); Betaine Hydrochloride (1500mg) PO x1 AND Ritonavir (100mg) PO x1 and Atazanavir (300mg) PO x1 on Day 4
  Arms: Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine HCl

SUMMARY:
The goal of this study is to evaluate the ability of a natural supplement (betaine hydrochloride) to affect the absorption of atazanavir in healthy volunteers. The investigators predict that betaine hydrochloride will increase the absorption of atazanavir in volunteers pre-treated with proton-pump inhibitors (PPIs).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age
* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam and laboratory evaluations
* BMI between 18.5-30 kg/m2
* Taking no medications 2 weeks before and during the study enrollment, including drugs of abuse, prescription or over-the-counter (OTC) medications (except acetaminophen)
* Subjects able to maintain adequate birth control during the study independent of hormonal contraceptive use
* Be able to provide written informed consent and comply with requirements of the study
* Avoid eating grapefruit and drinking grapefruit juice from 7 days before the first study day until the completion of the entire study
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 3pm the night before a study day until completion of that study day
* Fast from food and beverages at least 8 hours prior to medication dosing
* Be able to read, speak, and understand English

Exclusion Criteria:

* Subjects with a history of gastrointestinal disease including gastroesophageal reflux disease, gastritis, peptic ulcer disease, or dyspepsia
* Subjects with a fasting gastric pH of > 4 (i.e. hypochlorhydria)
* Subjects with a history of dysphagia, achalasia, or difficulty swallowing capsules, tablets, or pills
* Subjects on prescription or chronic over-the-counter (OTC) medications (including hormonal contraceptives)
* Subjects with known allergies rabeprazole, any other proton pump inhibitors (PPI's) or betaine hydrochloride
* Subjects who smoke tobacco
* Subjects with ongoing alcohol or illegal drug use
* Subjects who are pregnant, lactating, or attempting to conceive
* Subjects unable to maintain adequate birth control during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Area-Under-the Concentration Curve from zero-to-twenty two hours (AUC,0-22) of Atazanavir | Day 4
  The primary outcome measure will be atazanavir area-under-the-concentration curve (AUC) values from zero-to-twenty two (0-22) hours. Values from Experimental Arms of the study (Ritonavir-boosted Atazanavir plus Rabeprazole; Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine Hydrochloride) will be compared against the active comparator (Ritonavir-boosted atazanavir alone) and tested for statistical significance.
Area-Under-the Concentration Curve from zero-to-infinity (AUC,0-inf) of Atazanavir | Day 4
  The primary outcome measure will be atazanavir area-under-the-concentration curve (AUC) values from zero-to-infinite time (0-inf). Values from Experimental Arms of the study (Ritonavir-boosted Atazanavir plus Rabeprazole; Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine Hydrochloride) will be compared against the active comparator (Ritonavir-boosted Atazanavir alone) and tested for statistical significance.

SECONDARY OUTCOMES:
Maximum Concentration of Atazanavir | Day 4
  The maximum plasma concentration (Cmax) will also be measured. Values from Experimental Arms of the study (Ritonavir-boosted Atazanavir plus Rabeprazole; Ritonavir-boosted Atazanavir plus Rabeprazole AND Betaine Hydrochloride) will be compared against the active comparator (Ritonavir-boosted Atazanavir alone) and tested for statistical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, UCSF, San Francisco, California, United States